CLINICAL TRIAL: NCT00434967
Title: A Double-blind, Randomised, 4-arm Parallel Group, Multicentre, 8-week, Phase III Study to Assess the Antihypertensive Efficacy and Safety of the Combination of Candesartan Cilexetil (CC) 32 mg and Hydrochlorothiazide (HCT) 25 mg Compared With CC 32 mg, HCT 25 mg and Placebo in Hypertensive Adults
Brief Title: Antihypertensive Efficacy and Safety of Candesartan/HCT 32/25 mg in Comparison With Individual Components and Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2456C00002; EudraCT No. 2006-003963-30
Record Dates: First submitted 2007-02-13; First posted 2007-02-14 (Estimated); Results first posted 2009-06-17 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-11

CONDITIONS: Hypertension
Keywords: Blood pressure reduction; combination therapy; candesartan cilexetil; hydrochlorothiazide
MeSH Terms: conditions — Hypertension | interventions — candesartan cilexetil; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 4 (No Intervention): Placebo
- 2 (Active Comparator): Candesartan cilexetil
  Interventions: Drug: Candesartan cilexetil
- 3 (Active Comparator): Hydrochlorothiazide (HCT)
  Interventions: Drug: Hydrochlorothiazide
- 1 (Experimental): Candesartan cilexetil + Hydrochlorothiazide Combination
  Interventions: Drug: Candesartan cilexetil; Drug: Hydrochlorothiazide; Drug: Candesartan/HCT 32/25 mg

INTERVENTIONS:
Drug: Candesartan cilexetil — 32 mg oral tablet
  Other Names: ATACAND
  Arms: 1; 2
Drug: Hydrochlorothiazide — 25 mg oral tablet
  Other Names: HCTZ
  Arms: 1; 3
Drug: Candesartan/HCT 32/25 mg
  Arms: 1

SUMMARY:
The aim is to compare the blood pressure lowering effect of the combination of candesartan cilexetil (candesartan) 32 mg and hydrochlorothiazide (HCT) 25 mg to that of candesartan 32 mg alone, HCT 25 mg alone and placebo in hypertensive adults.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for enrolment into the study (Visit 1) if they fulfil all of the following criteria:
* Provision of signed Informed Consent
* Primary hypertension, untreated or treated with a maximum of 2 antihypertensive drugs (substances), which the patient and the physician are willing to withdraw at enrolment and replace with placebo.
* Mean sitting DBP 90-114 mmHg (value calculated in the eCRF) at Visits 1 and 2
* Patients will be eligible for randomisation (Visit 4) if they fulfil the following criterion:
* Mean sitting DBP of 90-114 mmHg (value calculated in the eCRF) at the end of the 4-week single-blind placebo run-in period. The run-in period should not be shorter than 4 weeks.

Exclusion Criteria:

* Pregnant or lactating women, or women of childbearing potential not practising an adequate method of contraception eg, intrauterine device, oral contraception or progesterone implant. Pregnancy must be excluded by a negative pregnancy test at Visit 1.
* Secondary or malignant hypertension
* Sitting SBP of 180 mmHg or more
* Myocardial infarction, stroke, coronary bypass surgery or transient ischaemic attack within 6 months before enrolment
* Angina pectoris requiring more treatment than short-acting nitrates
* Chronic use of NSAIDs
* Aortic or mitral valve stenosis
* Cardiac failure requiring treatment
* Cardiac arrhythmia requiring treatment
* Gout
* Renal artery stenosis or kidney transplantation
* Intravascular volume depletion
* Hypersensitivity to any component of the investigational products or to any sulphonamide derived drugs
* Concomitant disease which may interfere with the assessment of the patient
* Past or present alcohol or drug abuse, or any condition associated with poor compliance that in the opinion of the investigator might affect the patient's participation in the study
* Chronic liver disease
* Concomitant or previous treatment with any other investigational drug within 20 days of enrolment
* Previous enrolment in the present study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2207 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Klibaner, MD, Study Director — AstraZeneca; Istvan Edes, MD, Principal Investigator — DEOEC Institute of Cardiology
Locations (27):
- Belgium (8):
  - Research Site, Dour
  - Research Site, Gozée
  - Research Site, Hasselt
  - Research Site, Linkebeek
  - Research Site, Marchovelette
  - Research Site, Ronquières
  - Research Site, Saint-Médard
  - Research Site, Steenokkerzel
- Latvia (3):
  - Research Site, Daugavpils
  - Research Site, Ogre
  - Research Site, Riga
- Malta (2):
  - Research Site, Gozo
  - Research Site, Gwardiamangia
- Romania (7):
  - Research Site, Arad
  - Research Site, Bucharest
  - Research Site, Iași
  - Research Site, Piteşti
  - Research Site, Ploieşti
  - Research Site, Târgovişte
  - Research Site, Timișoara
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Slovakia (5):
  - Research Site, Bratislava
  - Research Site, Levice
  - Research Site, Lučenec
  - Research Site, Prešov
  - Research Site, Šahy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Following a screening evaluation, patients underwent a 4-week, single-blind treatment with placebo, after which eligible patients were randomly allocated in a 5:5:5:1 ratio to receive 8 weeks of double-blind treatment either with candesartan/Hydrochlorothiazide (HCT) 32/25 mg or candesartan 32 mg or HCT 25 mg or placebo, respectively.
Pre-assignment Details: In total, 2207 patients were enrolled in the study at 128 centres in 10 countries, 1772 patients received run in medication and 1524 patients were subsequently randomised to double-blind treatment.
Groups:
- Placebo: given as 2 placebo tablets corresponding to candesartan/HCT 16/12.5 mg tablets, 1 placebo tablet corresponding to a candesartan 32 mg tablet and 2 placebo tablets corresponding to HCT 12.5 mg tablets for double dummy blinding purpose)
- Candesartan 32 mg: candesartan 32 mg (given as 1 candesartan 32 mg tablet plus 2 placebo tablets corresponding to candesartan/Hydrochlorothiazide (HCT) 16/12.5 mg tablets and 2 placebo tablets corresponding to HCT 12.5 mg tablets for double dummy blinding purposes)
- HCT 25 mg: HCT 25 mg (given as 2 HCT 12.5 mg tablets plus 2 placebo tablets corresponding to candesartan/HCT 16/12.5 mg tablets and 1 placebo tablet corresponding to a candesartan 32 mg tablet for double dummy blinding purpose)
- Candesartan/HCT 32/25 mg: candesartan/HCT 32/25 mg (given as 2 candesartan/HCT 16/12.5 mg tablets, plus 1 placebo tablet corresponding to candesartan 32 mg tablet and 2 placebo tablets corresponding to HCT 12.5 mg tablets for double dummy blinding purposes)
Period: Overall Study
Arm/Group | Placebo | Candesartan 32 mg | HCT 25 mg | Candesartan/HCT 32/25 mg
Started | 97 | 465 | 470 | 492
Completed | 90 | 457 | 461 | 478
Not Completed | 7 | 8 | 9 | 14
Not completed — Adverse Event | 2 | 4 | 3 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 4 | 6
Not completed — Randomized in error | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 1
Not completed — Physician Decision | 1 | 1 | 1 | 0
Not completed — Patient Disposition Challenges | 2 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Candesartan 32 mg | HCT 25 mg | Candesartan/HCT 32/25 mg | Total
Number analyzed (Participants) | 92 | 457 | 464 | 486 | 1499
Age Continuous [Mean (Full Range); unit: years] | 52.7 [28 to 76] | 51.7 [21 to 79] | 50.9 [21 to 78] | 52.7 [22 to 77] | 52 [21 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 255 | 273 | 285 | 864
  Male | 41 | 202 | 191 | 201 | 635

OUTCOME MEASURES:

1. Primary Outcome: Change in Sitting Diastolic Blood Pressure (DBP) From Baseline to the End of the Study (From Baseline to 8 Weeks).
Description: Change (reduction) in sitting DBP at the end of the study, when compared to sitting DBP at baseline.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Candesartan 32 mg | HCT 25 mg | Candesartan/HCT 32/25 mg
Number analyzed (Participants) | 89 | 431 | 441 | 464
mm Hg | -3.3 (0.9) | -9.3 (0.4) | -7.7 (0.4) | -13.9 (0.4)

2. Primary Outcome: Change in Sitting Systolic Blood Pressure (SBP) From Baseline to the End of the Study (Baseline to 8 Weeks)
Description: Change (reduction) in sitting SBP at the end of the study, when compared to sitting SBP at baseline.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Candesartan 32 mg | HCT 25 mg | Candesartan/HCT 32/25 mg
Number analyzed (Participants) | 89 | 431 | 441 | 464
mm Hg | -3.7 (1.5) | -13.1 (0.7) | -11.6 (0.7) | -21.4 (0.6)

3. Secondary Outcome: The Number of Patients With Controlled Sitting DBP and Sitting SBP in Each Treatment Group at the End of the Study
Description: Controlled sitting SBP and sitting DBP are defined as having sitting SBP < 140 mmHg and sitting DBP < 90 mmHg at the end of the study
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Placebo | Candesartan 32 mg | HCT 25 mg | Candesartan/HCT 32/25 mg
Number analyzed (Participants) | 89 | 431 | 441 | 464
participants | 8 | 198 | 168 | 304

4. Secondary Outcome: Compare Candesartan/HCT 32/25 mg to Its Components and to Placebo With Regard to Hypertension Control Rate at the End of the Study (Patients With Controlled Sitting SBP and Sitting DBP).
Time Frame: Baseline to 8 weeks
Reporting Status: Not Posted

5. Secondary Outcome: To Describe Safety and Tolerability of the Study Treatments With Regard to Adverse Events Including Those That Lead to Treatment Discontinuation as Well as With Regard to Pulse Rate, Laboratory, Electrocardiographic and Physical Examination Findings.
Time Frame: Baseline to 8 weeks
Reporting Status: Not Posted

6. Secondary Outcome: To Compare Treatment With Candesartan/HCT 32/25 mg to Each of Its Components With Regard to Change From Baseline to Week 8 in Standing DBP and Standing SBP.
Time Frame: Baseline to 8 weeks
Reporting Status: Not Posted

7. Secondary Outcome: To Compare Candesartan/HCT 32/25 mg to Its Components and to Placebo With Regard to Sitting DBP Control Rate at the End of the Study (Patients With Controlled Sitting DBP Are Defined as Having a Sitting DBP <90 mmHg at the End of the Study).
Time Frame: Baseline to 8 weeks
Reporting Status: Not Posted

8. Secondary Outcome: To Compare Candesartan/HCT 32/25 mg to Its Components and to Placebo With Regard to Sitting DBP Responder Rate (Decrease in Sitting DBP ≥10 mmHg From Baseline to the End of the Study or a Sitting DBP <90 mmHg at the End of the Study).
Time Frame: Baseline to 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Placebo | Candesartan 32 mg | HCT 25 mg | Candesartan/HCT 32/25 mg
Serious Adverse Events (participants affected / at risk) | 2 | 6 | 2 | 1
Other Adverse Events (participants affected / at risk) | 0 | 38 | 22 | 23
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Placebo | Candesartan 32 mg | HCT 25 mg | Candesartan/HCT 32/25 mg
Acute Coronary Syndrome (Cardiac disorders) | 0/97 | 0/465 | 1/470 | 0/492
Back Pain (Musculoskeletal and connective tissue disorders) | 0/97 | 1/465 | 0/470 | 0/492
Cardiac Failure (Cardiac disorders) | 1/97 | 0/465 | 0/470 | 0/492
Cerebrovascular Accident (Nervous system disorders) | 0/97 | 1/465 | 0/470 | 0/492
Electrocardiogram Abnormal (Investigations) | 1/97 | 0/465 | 0/470 | 0/492
Hypotension (Cardiac disorders) | 0/97 | 0/465 | 0/470 | 1/492
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0/97 | 1/465 | 0/470 | 0/492
Major Depression (Psychiatric disorders) | 0/97 | 1/465 | 1/470 | 0/492
Pneumonia (Infections and infestations) | 0/97 | 1/465 | 0/470 | 0/492
Sudden Death (Infections and infestations) | 0/97 | 1/465 | 0/470 | 0/492
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Placebo | Candesartan 32 mg | HCT 25 mg | Candesartan/HCT 32/25 mg
Dizziness (Nervous system disorders) | 0/97 | 0/465 | 0/470 | 13/492
Headache (Nervous system disorders) | 0/97 | 18/465 | 22/470 | 10/492
Hypertension (Cardiac disorders) | 0/97 | 10/465 | 0/470 | 0/492
Influenza (Infections and infestations) | 0/97 | 10/465 | 0/470 | 0/492

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AstraZeneca shall have a period of 30 days from receipt of the proposed final manuscript for any publication or other disclosure to review it and may within such time require that submission for publication or disclosure of the manuscript be delayed in order for AstraZeneca to file patent applications.